CLINICAL TRIAL: NCT01789346
Title: Randomized, Controlled, Open-Label Pilot Study of a Novel 532 nm KTP Laser for the Treatment of Fresh Surgical Scars.
Brief Title: Pilot Study of a Novel 532nm KTP Laser for the Treatment of Fresh Surgical Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-12-EV03
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Scar; Surgical Scar; Cicatrix; Cicatrix, Hypertrophic; Keloid
Keywords: Scar; Scars; Surgical Scar; Surgical Scars; Cicatrix; Hypertrophic Cicatrix; Keloid; Hypertrophic Scar; Surgical Incision; Scarring; Abdominoplasty; Tummy Tuck; Augmentation Mammoplasty; Breast Augmentation; Thyroidectomy
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic; Keloid; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 532nm KTP (Other): Cutera ExcelV 532nm potassium titanyl phosphate (KTP) laser
  Interventions: Device: 532nm KTP
- 595nm PDL (Active Comparator): Cynosure Cynergy 595nm pulsed-dye (PDL) laser
  Interventions: Device: 595nm PDL

INTERVENTIONS:
Device: 532nm KTP — up to three treatments of 1/2 of Single scar, or one entire, randomized Bilateral scar.
  Other Names: ExcelV laser; Cutera ExcelV; Excel V
  Arms: 532nm KTP
Device: 595nm PDL — up to three treatments of 1/2 of Single scar, or one entire, randomized Bilateral scar.
  Other Names: Cynosure Cynergy; Cynergy laser
  Arms: 595nm PDL

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the 532nm potassium titanyl phosphate (KTP) laser in comparison with the 595nm pulsed-dye laser (PDL) for the treatment of fresh surgical scars.

DETAILED DESCRIPTION:
Randomized, Controlled, Open-Label Pilot Study of a Novel 532 nm KTP Laser for the Treatment of Fresh Surgical Scars. This is a single-center prospective, randomized, open-label, pilot study of a novel 532 nm KTP Laser in comparison with the 595nm pulsed-dye laser (PDL) in up to 20 subjects who have had a fresh surgical scar acquired within one to twelve months of the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I - IV
* Has postoperative linear scar(s) which is one to twelve months post-surgery.
* Having one scar that measures a minimum of 5 cm in length or two scars (bilateral) each measure a minimum of 2 cm in length.
* Be in good health.
* Must agree not to undergo any other procedure for the treatment of scar during the study.
* Willing to refrain from excess sun exposure and willing to wear sunscreen on the treated scar during the study (including the follow-up period).
* Able to read, understand and sign the Informed Consent Form.
* Willing and able to adhere to the treatment and follow-up schedule, and the post-treatment care instructions.
* Willingness to have digital photographs taken of the treated scar.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

* Participation in a study of another device or drug within 6 months prior to enrollment or during the study.
* Having received any prior treatment for the target surgical scar.
* Pregnant and/or breastfeeding.
* Significant concurrent illness, malignant tumors in the target area, acute or chronic skin infection/inflammation, currently using immunosuppressive medications or currently undergoing systemic chemotherapy.
* Current use of any medication known to increase sensitivity to light or taking prescription anticoagulation medication.
* History of abnormal or delayed wound healing, keloid formation or pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* History of malignant skin disease, immune deficiency disorders, coagulation disorders, seizure disorders due to light, or diseases stimulated by heat, unless prophylactic measures taken prior to treatment.
* Systemic use of isotretinoin within 6 months or corticosteroids within 12 months of study participation.
* Anytime in life, had used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Current smoker or history of smoking within 12 months of study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03-26 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Alster, MD, Principal Investigator — Washington Institute of Dermatologic Laser Surgery; Elizabeth Tanzi, MD, Principal Investigator — Washington Institute of Dermatologic Laser Surgery
Locations (1):
- Washington Institute of Dermatologic Laser Surgery, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Halves or single scars treated
Groups:
- All Study Participants: Patients with matched bilateral erythematous surgical scars or a single linear erythematous scar measuring longer than 5 cm were enrolled in the study. Single scars were divided into equal halves, with each half randomized to receive treatments with either a 532-nm KTP laser (Excel V; Brisbane, CA) or a 595-nm PDL (Cynergy; Cynosure Inc., Chelmsford, MA) at equivalent laser parameters. Bilateral matched scars were similarly randomized to receive 532-nm KTP or 595-nm PDL treatments.
Period: Overall Study
Arm/Group | All Study Participants
Started | 20; 40 Halves or single scars treated
Treatment With 532 nm KTP Laser | 20; 20 Halves or single scars treated
Treatment With 595 nm PDL Laser | 20; 20 Halves or single scars treated
Completed | 18; 36 Halves or single scars treated
Not Completed | 2; 4 Halves or single scars treated

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects treated with Cutera ExcelV 532nm KTP laser or Cynosure Cynergy 595nm pulsed-dye laser
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Surgical Scar of Treatment (532nm KTP Laser) and Active Control (595nm PDL) Treatment Arms.
Description: Improvement in surgical scar of 532 nm KTP and 595 nm PDL treatment arms at 12 weeks post-final treatment (compared to baseline) as assessed by blinded independent reviewers Physician's Global Assessment (min=0; max=3) Higher scores mean better outcome
Time Frame: 12-weeks post-final laser treatment
Measure: Median (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Halves or single scars treated
Groups:
- 532nm KTP Laser: Cutera ExcelV 532nm KTP laser
  532nm potassium titanyl phosphate (KTP) laser
- 595nm PDL: Cynosure Cynergy 595nm pulsed-dye laser
  595nm pulsed-dye laser (PDL)
Arm/Group | 532nm KTP Laser | 595nm PDL
Number analyzed (Participants) | 18 | 18
Number analyzed (Halves or single scars treated) | 18 | 18
score on a scale | 2.0 [1.0 to 2.5] | 1.5 [0.0 to 2.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first laser treatment through completion of the study for all subjects (24 weeks)
Description: Systematic assessment occurred through regular investigator assessments during study visits. Between visits, participants were also encouraged to contact the site to report any adverse events that occurred as applicable.
Arm/Group | 532nm KTP Laser | 595nm PDL
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 532nm KTP Laser (N=19) | 595nm PDL (N=19)
Erythema (Skin and subcutaneous tissue disorders) | 9 | 7
Edema (Skin and subcutaneous tissue disorders) | 2 | 2
Purpura (Skin and subcutaneous tissue disorders) | 3 | 1
Crusting (Skin and subcutaneous tissue disorders) | 2 | 0
Burning Sensation (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No